CLINICAL TRIAL: NCT01590836
Title: A Trial Investigating the Pharmacodynamic Properties of NN5401 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1979; 2011-003797-90 (EudraCT Number); U1111-1123-3837 (Other: WHO)
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDeg-->IDegAsp (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Administered subcutaneously (s.c., under the skin) once daily (plus insulin aspart as bolus insulin as required).
Drug: insulin degludec/insulin aspart — Single dose administered subcutaneously (s.c., under the skin).

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacodynamic response (the effect of the investigated drug on the body) of insulin degludec/insulin aspart (IDegAsp) at steady state in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for at least 12 months
* Body mass index (BMI) 18.0-28.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin (HbA1c) maximum 9.5 %
* Fasting C-peptide maximum 0.3 nmol/L

Exclusion Criteria:

* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking, use of nicotine gum or transdermal nicotine patches during the inpatient period
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Surgery or trauma with significant blood loss (more than 500 mL) within the last 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval | At steady state (0-24 hours)

SECONDARY OUTCOMES:
Maximum glucose infusion rate (GIRmax) | At steady state (within 0-24 hours after last dosing)
Area under the serum insulin degludec concentration-time curve during one dosing interval | At steady state (within 0-24 hours after last dosing)
Maximum observed serum insulin degludec concentration | At steady state (within 0-24 hours after last dosing)
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours
Maximum observed serum insulin aspart concentration | Within 0-12 hours after dosing of IDegAsp

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Nosek L, Roepstorff C, Chenji S, Klein O, Haahr H. Distinct Prandial and Basal Glucose-Lowering Effects of Insulin Degludec/Insulin Aspart (IDegAsp) at Steady State in Subjects with Type 1 Diabetes Mellitus. Diabetes Ther. 2014 Jun;5(1):255-65. doi: 10.1007/s13300-014-0070-2. Epub 2014 Jun 3. PMID 24888255
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com